CLINICAL TRIAL: NCT05901805
Title: Validation of the Occupational Sitting and Physical Activity Questionnaire for E-Sports Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc. Prof. Dr., Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC2023
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Physical Inactivity; Sedentary Time; Pain
Keywords: Gaming; Esport; Questionnaire; physical activity
MeSH Terms: conditions — Sedentary Behavior; Pain; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire application — Participants will be asked to fill in the "Occupational Sitting and Physical Activity Questionnaire" adapted into Turkish. Correlation of the scale with the International Physical Activity Questionnaire-Short Form, VAS and YİBT-SF, Buss-Perry Aggression Scale will be tested. The questionnaire will be repeated every 7-14 days in order to perform the test-retest analysis of the questionnaire.

SUMMARY:
Electronic sports (Esports) has become a branch that started to gain popularity in the gaming community in the early 2000s and that more and more individuals are interested in. Esports players are often called sedentary athletes because gaming requires prolonged sedentary activity. The aim of this study is to adapt the Occupational Sitting and Physical Activity Questionnaire to individuals playing Esports and to validate it in Turkish.

DETAILED DESCRIPTION:
Electronic sports (Esports) has become a branch that started to gain popularity in the gaming community in the early 2000s and that more and more individuals are interested in. Esports players are often called sedentary athletes because gaming requires prolonged sedentary activity. Although studies have examined the physical activity levels of Esports players with questionnaires, they emphasize that the results may be more variable because they do not control for potential confounding factors such as gender, age, game type, and performance level. Among the questionnaires used in the studies, there was no study evaluating the player-specific physical activity level. Therefore, the aim of this study is to validate the Occupational Sitting and Physical Activity Questionnaire in individuals playing Esports. Individuals aged 12-24, who play computer games 3-4 times a week for 2-4 hours professionally or 7-14 hours a week as an amateur, and have the ability to read and understand Turkish will be included in the study. Individuals with severe physical limitations that prevent physical activity and individuals with cognitive impairment will be excluded from the study. Correlation of the scale with Visual Analogue Scale (VAS), International Physical Activity Questionnaire-Short Form for construct validity, Young Internet Addiction Test-Short Form (YİBT-SF) and Buss-Perry Aggression Scale will be tested, respectively. In order to determine the test-retest reliability of the Turkish version of the scale, individuals will be asked to fill in the scale again 7-14 days after they first filled out the scale.

ELIGIBILITY:
Inclusion Criteria:

ESports Players:

* Volunteer to participate in the study
* Age between of 12-24
* Training for 2-4 hours 3-4 times a week
* Playing e-sports for at least 1 year
* Play and be licensed as an active esports player in an official esports tournament or league

Amateur Recreational players:

* Not having an e-athlete license
* Age between of 12-24
* Playing games 7-14 hours a week
* Have an active game account in any region

Exclusion Criteria:

ESports Players:

* Having had a head injury accident within the last week
* No e-sports license
* Having a congenital disease or deformity
* Having a diagnosis of psychiatric and neurological disease
* Having a diagnosis of musculoskeletal disease

Amateur Recreational players:

* Having a systemic or congenital disease
* Having a diagnosis of neurological and psychiatric disease
* Having a disorder that affects the musculoskeletal system

Ages: 12 Years to 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: Esports and amateur recreational players between the ages of 12-24 who agree to voluntarily participate in the study will be included.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Occupational Sitting and Physical Activity Questionnaire (OSPAQ) | Baseline (First assessment)
  Occupational Sitting and Physical Activity Questionnaire; It is a short scale that records the proportion of working time spent sitting, standing, walking, and doing heavy work, and the total time worked in the last five working days. Participants will be asked to indicate the percentage of time they spend on these activities in a day. All percentages specified by participants for sitting, standing, walking and heavy work activities will be added up.

SECONDARY OUTCOMES:
Occupational Sitting and Physical Activity Questionnaire (OSPAQ) | Within a 7-to-14-day period after the first assessment (Second assessment)
  Occupational Sitting and Physical Activity Questionnaire; It is a short scale that records the proportion of working time spent sitting, standing, walking, and doing heavy work, and the total time worked in the last five working days. Participants will be asked to indicate the percentage of time they spend on these activities in a day. All percentages specified by participants for sitting, standing, walking and heavy work activities will be added up.
International Physical Activity Questionnaire-Short Form (IPAQ-Short Form) | Baseline (First assessment)
  IPAQ was developed to measure the health and physical activity levels of the society. This global scale allows the assessment of physical activity. The short version provides information about the time spent walking, moderate and vigorous activities, and sedentary activities. Outcome evaluation is carried out by reporting weekly activity duration with an estimation of MET energy expenditure for each activity category.
Visual Analogue Scale (VAS) | Baseline (First assessment)
  The VAS is a pain assessment scale using a 10 cm line graded as "no pain" 0 points and "worst pain imaginable" 10 points.
Young Internet Addiction Test-Short Form (YİBT-SF) | Baseline (First assessment)
  The YİBT-SF, which measures internet addiction, consists of 12 items and is a five-point Likert scale (1=Never, 5=Very often).
Buss-Perry Aggression Questionnaire | Baseline (First assessment)
  It is an aggression assessment scale consisting of 34 items. The situations described in the items question five sub-forms of aggression (physical aggression, verbal aggression, anger, hostility, and indirect aggression). It is a five-point Likert-type self-rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided